CLINICAL TRIAL: NCT05768165
Title: Expected Health Benefits on Cardiovascular Function, Inflammation and Quality of Life With High-intensity Interval Exercise for Patients With Rheumatoid Arthritis
Brief Title: High-intensity Interval Exercise in Rheumatoid Arthritis
Acronym: RA-HIIT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vastra Gotaland record 275642
Record Dates: First submitted 2021-09-06; First posted 2023-03-14 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Intervention versus care as usual
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Cardiorespiratory and strength exercise training 2-3 sessions per week
  Interventions: Behavioral: High intensity exercise
- Care as usual (No Intervention): Care as usual and information of health enhancing physical activity according to general recommendations

INTERVENTIONS:
Behavioral: High intensity exercise — Twelve weeks of supervised high intensity aerobic and resistance exercise including two sessions/week, one additional session of the patient´s own choice, non-supervised. The target of the high intensity intervals (HIIT) is 90%-95% of maximum heart rate alternated with recovery phases at 70% of maximal heart rate. The resistance exercise session of large muscle groups: 8-10 repetitions, 2-3 sets.
  Exercise guidance follows principles of self-efficacy and person-centeredness.
  Other Names: Person- centeredness
  Arms: Intervention group

SUMMARY:
Cardiovascular performance and overall fitness can be improved by high-intensity aerobic activity, and these benefits may be achievable by persons with rheumatic diseases. The investigators hypothesize that a 12-week high-intensity interval exercise program will provide substantial improvements in cardiovascular function, inflammation and symptoms affecting quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis disease according to the American College of Rheumatology (ACR)/ The European Alliance of Associations for Rheumatology (EULAR) 1987/2010 criteria
* Disease duration >1 year
* Age (range 20-60 years)
* Stable medication on anti- rheumatic drugs for >3 months
* Low-to-moderate disease activity (<5.1) according to the Disease activity score 28 (DAS28)

Exclusion Criteria:

* Cerebrovascular diseases
* Diabetes
* Severe hypertension
* Chronic obstructive pulmonary disease or other severe pulmonary diseases
* Other severe diseases that may be associated with adverse events or restrict participation in high-intensity exercise
* Arthroplasty of large joints
* Inability to manage Cardiopulmonary Exercise Testing (CPET)
* Pregnancy
* Already participating in regular aerobic or strength exercise at a high intensity level (>1 hours/ week) during the last 6 months
* Inability to speak or read Swedish.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary function | 0 -12 weeks
  Maximum oxygen uptake (VO2ml/min/kg) (Higher value indicate better cardiorespiratory capacity)

SECONDARY OUTCOMES:
Vascular function | 0-12 weeks
  Aortic pulse wave velocity (PWV) (m/sec.) (Higher PWV value indicate worse vascular function)
Level of disease activity | 0-12 weeks
  Disease activity score 28 (DAS28) (Range 0-10 where a higher score indicate worse disease activity)
Level of disease activity | 0-6 months
  Disease activity score 28 (DAS28) (Range 0-10 where a higher score indicate worse disease activity)
Level of disease activity | 0-12 months
  Disease activity score 28 (DAS28) (Range 0-10 where a higher score indicate worse disease activity)
Homeostatic model assessment of insulin resistance (HOMA IR) | 0-12 weeks
  Measure of insulin resistance (fasting glucose (mmol/L) and fasting insulin (mIU/ L) will be combined to report HOMA IR
Glycosylation level of hemoglobin (HbA1c) | 0-12 weeks
  Glycosylation level of hemoglobin (mmol/mol)
Level of blood lipids | 0-12 weeks
  Levels of triglycerides (mmol/L), Level of high-density lipoprotein (HDL) (mmol/L), low-density lipoprotein (LDL) ( mmol/L), Total cholesterol (mmol/L )
Erythrocyte Sedimentation Rate (ESR) | 0-12 weeks
  Level of high sensitivity ESR (mm/h) (Higher score indicate higher inflammation)
Erythrocyte Sedimentation Rate (ESR) | 0-6 months
  Level of high sensitivity ESR (mm/h) (Higher score indicate higher inflammation)
Erythrocyte Sedimentation Rate (ESR) | 0-12 months
  Level of high sensitivity ESR (mm/h) (Higher score indicate higher inflammation)
C-Reactive Protein (CRP) | 0-12 weeks
  Level of high sensitivity CRP (mg/L) (Higher score indicate higher inflammation)
C-Reactive Protein (CRP) | 0-6 months
  Level of high sensitivity CRP (mg/L) (Higher score indicate higher inflammation)
C-Reactive Protein (CRP) | 0-12 months
  Level of high sensitivity CRP (mg/L) (Higher score indicate higher inflammation)
Cytokine levels | 0-12 weeks
  Interleukin-6 (pg/mL), interleukin-10 (pg/mL), tumour necrosis factor-alpha (pg/mL)
Muscle function of lower extremities | 0-12 weeks
  The one minute sit-to-stand test (Higher numbers of complete rises indicate better muscle function in lower extremities)
Hand-grip force | 0-12 weeks
  Hand-grip force is assessed with a dynamometer ( Higher value indicate better grip strength)
Self-reported physical activity | 0-12 weeks
  Self-reported questionnaire of habitual physical activity during a typical week. Numbers of hours on low, moderate and high intensity is summed for each category (A minimum of 150 minutes on moderate intensity or 75 minutes on high intensity are equal to health enhancing physical activity according to World Health Organization guidelines)
Self-reported physical activity | 0-6 months
  Self-reported questionnaire of habitual physical activity during a typical week. Numbers of hours on low, moderate and high intensity is summed for each category (A minimum of 150 minutes on moderate intensity or 75 minutes on high intensity are equal to health enhancing physical activity according to World Health Organization guidelines)
Self-reported physical activity | 0-12 months
  Self-reported questionnaire of habitual physical activity during a typical week. Numbers of hours on low, moderate and high intensity is summed for each category (A minimum of 150 minutes on moderate intensity or 75 minutes on high intensity are equal to health enhancing physical activity according to World Health Organization guidelines)
Objective assessment of physical activity | 0-12 weeks
  Accelerometer to assess habitual physical activity during a typical week. Total time of physical activity and physical activity pattern assessed as time spent at different physical activity intensity levels are obtained using the metabolic equivalent of task values (METS). (Higher METs value indicate higher physical activity level.)
Objective assessment of physical activity | 0-6 months
  Accelerometer to assess habitual physical activity during a typical week. Total time of physical activity and physical activity pattern assessed as time spent at different physical activity intensity levels are obtained using the metabolic equivalent of task values (METS). (Higher METs value indicate higher physical activity level.)
Objective assessment of physical activity | 0-12 months
  Accelerometer to assess habitual physical activity during a typical week. Total time of physical activity and physical activity pattern assessed as time spent at different physical activity intensity levels are obtained using the metabolic equivalent of task values (METS). (Higher METs value indicate higher physical activity level.)
Pain intensity | 0-12 weeks
  Visual Analogue Scale (VAS) (0-100, Higher score indicate worse pain)
Pain intensity | 0-6 months
  Visual Analogue Scale (VAS) (0-100, Higher score indicate worse pain)
Pain intensity | 0-12 months
  Visual Analogue Scale (VAS) (0-100, Higher score indicate worse pain)
Global health | 0-12 weeks
  Visual Analogue Scale (VAS) (0-100, Higher score indicate worse health)
Global health | 0-6 months
  Visual Analogue Scale (VAS) (0-100, Higher score indicate worse health)
Global health | 0-12 months
  Visual Analogue Scale (VAS) (0-100, Higher score indicate worse health)
Fatigue | 0-12 weeks
  The Multiple Fatigue Inventory (MFI-20) (4-20 for each subscale, Higher score indicates a higher degree of fatigue
Fatigue | 0-6 months
  The Multiple Fatigue Inventory (MFI-20) (4-20 for each subscale, Higher score indicates a higher degree of fatigue
Fatigue | 0-12 months
  The Multiple Fatigue Inventory (MFI-20) (4-20 for each subscale, Higher score indicates a higher degree of fatigue
Sleep | 0-12 weeks
  Pittsburgh Sleep Quality Index (0-21, Higher score indicate worse sleep quality).
Sleep | 0-6 months
  Pittsburgh Sleep Quality Index (0-21, Higher score indicate worse sleep quality).
Sleep | 0-12 months
  Pittsburgh Sleep Quality Index (0-21, Higher score indicate worse sleep quality).
Activity limitations | 0-12 weeks
  Health Assessment Questionnaire (HAQ) (0-3, Higher score indicate worse activity limitations)
Activity limitations | 0-6 months
  Health Assessment Questionnaire (HAQ) (0-3, Higher score indicate worse activity limitations)
Activity limitations | 0-12 months
  Health Assessment Questionnaire (HAQ) (0-3, Higher score indicate worse activity limitations)
Attitude to exercise | 0-12 weeks
  Exercise Health Beliefs questionnaire (20-100, Higher score represents stronger exercise health beliefs.
Attitude to exercise | 0-6 moths
  Exercise Health Beliefs questionnaire (20-100, Higher score represents stronger exercise health beliefs.
Attitude to exercise | 0-12 months
  Exercise Health Beliefs questionnaire (20-100, Higher score represents stronger exercise health beliefs.
Body compositions | 0-12 weeks
  Weight and height will be combined to report Body mass index BMI kg/m2 (A higher score indicate higher relative weight)
Waist circumference | 0-12 weeks
  Measured with a tape measure midway between the lower rib and iliac crest. (A waist measurement of 80 centimeters or more for women and 94 centimeters or more for men indicate increased risk for diseases related to overweight)

CONTACTS AND LOCATIONS:
Overall Officials: Annelie Bilberg, PhD, Study Director — Vastra Gotaland Region
Locations (2):
- Sweden (2):
  - Sahlgrenska university hospital, Gothenburg
  - Uddevalla Hospital, Uddevalla

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in a publication are available from the principal investigator (P.I.) on reasonable request. Access will be determined based on reasonable request and in accordance with the ethical approval
Time Frame: The data will become available as following, starting 6 months after publication and end 5 years after publication.
Access Criteria: The requests will be reviewed by the P.I. and the steering committee. Study plans on meta-analyses generating new knowledge on exercise in persons with rheumatic diseases will be approved.

REFERENCES:
- [Derived] Bilberg A, Bjersing J, Borjesson M, Sivertsson J, Mannerkorpi K. High-intensity exercise improves multidimensional fatigue and health-related quality of life in rheumatoid arthritis: a randomized controlled study. Arthritis Res Ther. 2025 Sep 18;27(1):176. doi: 10.1186/s13075-025-03643-3. PMID 40968365
- [Derived] Bilberg A, Mannerkorpi K, Borjesson M, Svedlund S, Sivertsson J, Klingberg E, Bjersing J. High-intensity interval training improves cardiovascular and physical health in patients with rheumatoid arthritis: a multicentre randomised controlled trial. Br J Sports Med. 2024 Dec 2;58(23):1409-1418. doi: 10.1136/bjsports-2024-108369. PMID 39179363